CLINICAL TRIAL: NCT04300985
Title: Magnesium Sulfate Versus Dexmedetomidine on Anesthesia Awakening. Randomized Clinical Trial.
Brief Title: Magnesium Sulfate Versus Dexmedetomidine on Anesthesia Awakening.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Associate professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE 28455419.9.0000.5448
Record Dates: First submitted 2020-02-29; First posted 2020-03-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Cholecystectomy
MeSH Terms: interventions — Dexmedetomidine; Anesthesia, General; Saline Solution; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: This is a prospective, controlled, blinded trial with random distribution.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One professional of the team of providers will be responsible for conducting the electronic drawing on the website www.random.org, to distribute 90 numbers randomly into three groups. By following the results he or she will identify 90 opaque envelopes with numbers, and inside of each envelope will be a card with the name of corresponding group and the instructions about the corresponding intervention. This professional will not take part in any other part of the investigation. Every other professionals of the team and the patient will be blinded to group to which the patient belong. Each of the invited patient who accepts to participate and sign the consent form in the pre-anesthetic consultation, will receive the sequential envelope and be part of the corresponding group. At the arrival in the surgical center, one particular professional of the team will open the envelope and prepare the blinded solution, that will still be unclosed to any other people in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Sham Comparator): Thirty patients in this group will receive infusion of 100 saline solution. After 15 min of beginning of this infusion they will start receiving general anesthesia administration.
  Interventions: Drug: Sham treatment
- Dexmedetomidine group (Active Comparator): Thirty patients in this group will receive infusion of dexmedetomidine (0,5 mcg/kg/min). After 15 min of the beginning of this infusion they will start in the general anesthesia induction.
  Interventions: Drug: Dexmedetomidine
- Magnesium sulfate group (Active Comparator): Thirty patients in this group will receive infusion of magnesium sulfate (20 mg/kg/h). After 15 min of the beginning of this infusion they will start in the general anesthesia induction.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will start receiving dexmedetomidine 15 minutes before general anesthetic induction.
  Other Names: Dexmedetomidine and general anesthesia
  Arms: Dexmedetomidine group
Drug: Sham treatment — Patients will start receiving saline solution infusion 15 minutes before general anesthetic induction.
  Other Names: Saline solution and general anesthesia
  Arms: Placebo group
Drug: Magnesium Sulfate — Patient will start receiving magnesium infusion (20 mg/kg/h) 15 minutes before general anesthetic induction.
  Other Names: Magnesium sulfate and general anesthesia
  Arms: Magnesium sulfate group

SUMMARY:
Magnesium sulfate (MS) and dexmedetomidine have already demonstrated the ability to reduce intra and postoperative consumption of anesthetics and analgesics, among others advantages, such as blood pressure control and intraoperative bleeding. The MS has also been shown to be useful in pre-eclampsia and eclampsia control, pulmonary hypertension, asthma, cardiac arrhythmias and pheochromocytoma). Despite these advantages in the use of these important adjuncts, there is a concern about the quality and awakening time of the patients who use them. The purpose of this trial is to compare the time and quality of awakening in patients submitted to general anesthesia and receiving MS or dexmedetomidine as adjuncts in the intraoperative analgesia.

The main objective of this trial is to compare the quality and the awakening time in patients receiving MS or dexmedetomidine. The secondary objective is the comparison of postoperative analgesia in the postoperative hospitalization period. Hypothesis: Our hypothesis is that patients present a faster awakening when receive MS as an analgesic adjunct, when compared to patients who receive dexmedetomidine. Drawing: this is a prospective, controlled, covert trial with random distribution for noninferiority trialing.

DETAILED DESCRIPTION:
INTRODUCTION Magnesium sulfate (MS) and dexmedetomidine have already demonstrated the ability to reduce intra and postoperative consumption of anesthetics and analgesics, among others advantages, such as blood pressure control and intraoperative bleeding8,9. The MS has also been shown to be useful in pre-eclampsia and eclampsia control, pulmonary hypertension, asthma, cardiac arrhythmias and pheochromocytoma). Despite these advantages in the use of these important adjuncts, there is a concern about the quality and awakening time of the patients who use them. The purpose of this trial is to compare the time and quality of awakening in patients submitted to general anesthesia and receiving MS or dexmedetomidine as adjuncts in the intraoperative analgesia.

The main objective of this trial is to compare the quality and the awakening time in patients receiving MS or dexmedetomidine. The secondary objective is the comparison of postoperative analgesia in the postoperative hospitalization period. Our hypothesis is that patients present a faster awakening when receive MS an analgesic adjunct, when compared to patients who receive dexmedetomidine.

Drawing: this is a prospective, controlled, covert trial with random distribution for noninferiority trialing.

Key words: general anesthesia, long awakening from anesthesia. METHODS Participants and endpoints Scenario: The study will be carried out at "Hospital da Sociedade Portuguesa de Beneficência de Santos - Angiocorpore" (Portuguese Charity Society Hospital). Eligibility: Patients scheduled for video laparoscopic cholecystectomy, between 18 and 70 years old, physical status I or II in the American Society of Anesthesiology classification, who have no allergy or contraindication to the study protocol substances and who voluntarily agree to participate in the trial and sign the informed consent form (TCLE), will be invited to participate in the study.

Coronary disease patients, patients with heart block > atrioventricular block > I, patients with renal failure, those with brain disease past history, dementia or other psychiatric diseases, and patients with body mass index > 35 kg/m², will be excluded. Also excluded patients with Portuguese language limitations and in preoperative use of opioid or corticosteroids.

Intervention: the sample of participants will be distributed in 3 groups. The placebo group (GP) will receive 100 ml of saline solution (SL) in infusion pump (BI) starting 15 min before anesthesia with flow of 0.25 ml/kg/h. The dexmedetomidine group (GD) will receive 100 ml of SL with 200 µg of dexmedetomidine in BI, starting 15 min before anesthesia with flow of 0.25 ml/kg/h. The magnesium sulfate group (GM) will receive 80 ml of MS + 20 ml of SL in infusion pump starting 15 min before anesthesia induction with flow of 0.25 ml/kg/h. With this infusion flow, patients of GD will receive dexmedetomidine at a dose of 0.5 µg/kg/h and patients of GM will receive MS at a dose of 20 mg/kg/h. All participants will be submitted to balanced anesthesia.

Anesthetic induction will be initiated after 5 min of pre-oxygenation, with lidocaine 1.5 mg/kg, fentanyl 3 µg/kg, propofol up to clinical hypnosis, cisatracurium 0.1 mg/kg and intubation after adequate neuromuscular relaxation. Maintenance will be with sevoflurane at a concentration under clinical demand, repeating bolus of fentanyl 1µg/kg and cisatracurium 0.03 mg/kg as needed.

Primary endpoints: time between the end of anesthetic administration and bispectral index > 60, and a battery of neuropsychological trials for evaluation of postoperative cognitive dysfunction tested in the Brazilian population 3 h after the end of anesthetics administration.

. Secondary endpoints: response to the questionnaire of the brief pain inventory and opioid consumption in the first 2 days of postoperative. Recruitment: patients will be recruited in the pre-anesthetic evaluation and the evaluations will be done in a covert way in the immediate postoperative period and during the two postoperative days, being recorded the pain scores and consumption of opioids.

Sample calculation: the sample of 73 participants was calculated for a 95% confidence index and a 90% statistical power. For compensation for losses, 90 individuals will be recruited distributed in 3 groups.

Recruitment and allocation Distribution in groups: through electronic drawing on the website www.random.org and preparation of brown envelopes that will be numbered and will contain inside a card with the name of the group to which that number corresponds, in addition to the intervention concerning the group to which it belongs. The draw and preparation of the envelopes will be conducted by a professional who will not participate in other stages of the study.

Masking: participants, providers and evaluators will be blinded to group each patient belongs to. The randomization and allocation will be performed by professional not participating in any other step of the trial.

Data collection and management Collection: the time between the end of anesthetic administration and bispectral index > 60 monitoring will be recorded; cognitive evaluation will be done at recruitment and 3 h after the end of the anesthesia; the brief pain inventory questionnaire will be filled in at recruitment and 3 h after the end of the anesthesia; during hospitalization and in the first 2 days of postoperative the opioid consumption will be registered.

Data management: the data will be organized in MS Excel spreadsheet, in its MS-Office 2013 version. The results will be obtained through the Statistical Package for Social Sciences (SPSS) in its version 23.0.

Statistical analysis: continuous variables will be evaluated through Student's t trial. The normality check will be evaluated by Kolmogorov-Smirnov trial or Shapiro-Wilk trial. The comparison of parametric data will be done by Student's t trial or Z trial. The nominal variables will be evaluated by the Chi-square trial. The comparison of nominal variables for independent samples will be made by the Chi-square trial or Fisher's Exact trial. The comparison of ordinal or quantitative variables without normal distribution for independent samples will be done by the Mann-Whitney trial. The correlation between variables will be evaluated by Pearson's trial for or Spearman, as indicated.

Patient follow-up The compared substances are already widely used in anesthesia and present a very favorable risk/benefit ratio, with no significant incidence of intercurrence related to them being noted. The selection of patients for the study also makes their use safe. To make the benefit of its use uniform among the groups, patients with pain scores > 3 (pain verbal score 0 to 10) will receive 2 mg of morphine at 15-minute intervals, until the pain intensity is < 3.

Participants will receive a prescription for home use of dipyrone 1g every 6 hours and association of codeine (30 mg) with paracetamol (500 mg) in case of pain > 3. RESEARCH ETHICS This project was submitted to the evaluation of the Research Ethics Committee (CEP/CONEP) in the Brazil Platform and to the Ethics Committee of participating institution. After their approval, it is being registered at clinicaltrials.org. Only after these steps the data collection will started.

The recruited individuals will only participate in the study after signing the consent form.

Participants' personal information will be kept confidential, and only the authors will have access to them before, during and after the trial. The authors declare that they have no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for video laparoscopic cholecystectomy, between 18 and 70 years old, physical status I ou II in the American Society of Anesthesiology classification

Exclusion Criteria:

* Allergy or contraindication to the study protocol substances, refuse to participate or sign the informed consent, heart block > atrioventricular I, renal failure, brain disease, dementia or other psychiatric diseases, body mass index > 35 kg/m², Portuguese language limitations, preoperative use of opioid or corticosteroids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Time to awake from anesthesia between groups | Three hours
  Comparing time in minutes to get bispectral index higher than 60 in both groups

SECONDARY OUTCOMES:
Comparing postoperative analgesia between groups | Two days
  Comparing opioid consumption in milligrams between groups

CONTACTS AND LOCATIONS:
Overall Officials: Sebastião Silva Filho, Principal Investigator — Hospital da Sociedade de Beneficência Portuguesa d
Locations (1):
- Hospital das Clínicas - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We may only share data related to exams, outcomes and other related with the trial, not personal information.

REFERENCES:
- [Background] 1. Telci L, Esen F, Akcora D, Erden T, Canbolat AT, Akpir K. Evaluation of effects of magnesium sulfate in reducing intraoperative anaesthetic requirements. Br J Anaesth. 2002; 89: 594-598. 2. Chen C, Tao R. The impact of magnesium sulfate on pain control after laparoscopic cholecystectomy: a meta-analysis of randomized controlled studies. Surg Laparosc Endosc Percutan. 2018; 28: 349-353. 3. Andjelkovic L, Novak-Jankovic V, Pozar-Lukanovic N, Bosnic Z, Spindler-Vesel A. Influence of dexmedetomidine and lidocaine on perioperative opioid consumption in laparoscopic intrialine resection: a randomized controlled clinical trial. J Int Med Res. 2018; 46: 5143-5154.